CLINICAL TRIAL: NCT07037134
Title: Impact of Auditory Environments on the Functioning of Pain Mechanisms in Fibromyalgia Syndrome: a Randomized, Triple-blind, Placebo-controlled 4×4 Crossover Trial
Brief Title: Impact of Auditory Environments on Pain in Fibromyalgia: a 4×4 Crossover Trial
Acronym: SoundsPainFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Associate Professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FIBRO-PAIN-SOUND-2025
Record Dates: First submitted 2025-06-09; First posted 2025-06-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia Syndrome
Keywords: Acoustic environment; Audioanalgesia; Blank tape; Broadband noise; Chronic primary pain; Clinical trial; Crossover; Fibromyalgia; Natural sound; Pain modulation; Pink noise; Soundscape; Urban sound; White noise
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study employs a randomized, triple-blind, placebo-controlled crossover design based on a 4×4 Williams Latin square. Each participant receives all four interventions in a randomized, balanced sequence across four periods, with one-week washout intervals separating each session to mitigate residual effects. The design ensures equal representation of each condition across periods and sequences (uniform within sequences and periods), controlling for first-order carryover effects. This model supports within-subject comparisons, minimizes interindividual variability and confounding, and improves statistical power and internal validity using robust outcome analysis via mixed-effects modeling.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a triple-blind design: intervention administrator, outcome assessor, and data analyst will be fully masked, while participants will remain unaware (masked, not blinded) of the study hypotheses. The intervention administrator will be blinded to the audio content being delivered, as stimuli will be labeled with non-descriptive codes by a separate investigator. The outcome assessor will not be involved in the intervention and will be blinded to group allocation. Participants will be instructed not to disclose any intervention-related information. Any potentially unblinding data that could reveal group allocation will be masked before it reaches the outcome assessor. The data analyst will receive fully de-identified datasets, with groups labeled only as "Group A/B/C/D"; unblinding will occur only after all analyses have been completed and verified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence NBPU (Other): Participants assigned to this sequence receive natural soundscape exposure in Week 1, broadband sound exposure in Week 2, placebo control (blank tape) in Week 3, and urban soundscape exposure in Week 4. Each session lasts 20 minutes, with one-week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound exposure; Other: Blank tape attention placebo control
- Sequence UPBN (Other): Participants assigned to this sequence receive urban soundscape exposure in Week 1, placebo control (blank tape) in Week 2, broadband sound exposure in Week 3, and natural soundscape exposure in Week 4. Each session lasts 20 minutes, with one week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound exposure; Other: Blank tape attention placebo control
- Sequence BUNP (Other): Participants assigned to this sequence receive broadband sound exposure in Week 1, urban soundscape exposure in Week 2, natural soundscape exposure in Week 3, and placebo control (blank tape) in Week 4. Each session lasts 20 minutes, with one week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound exposure; Other: Blank tape attention placebo control
- Sequence PNUB (Other): Participants assigned to this sequence receive placebo control (blank tape) in Week 1, natural soundscape exposure in Week 2, urban soundscape exposure in Week 3, and broadband sound exposure in Week 4. Each session lasts 20 minutes, with one week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound exposure; Other: Blank tape attention placebo control

INTERVENTIONS:
Other: Natural soundscape exposure — Participants receive a standardized 20-minute auditory exposure to curated natural soundscapes via high-fidelity open-back reference headphones powered by a DAC/amplifier and corrected for frequency response using calibration software. Participants are randomly assigned one of 22 recordings. Each includes 10-second fade-in/out effects and is calibrated to 45-55 dB. The stereo recordings (320-kbps MP3, 48 kHz/24-bit) feature biophony (e.g., bird vocalizations) and geophony (e.g., rainfall), free of urban sounds and selected for ecological validity based on predefined criteria: (i) recognizable/context-specific sounds; (ii) culturally neutral; (iii) foreground presence and depth; (iv) no prolonged silence; (v) no technical artifacts. During exposure, they lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening under continuous researcher supervision.
  Other Names: Experimental intervention N
Other: Urban soundscape exposure — Participants receive a standardized 20-minute auditory exposure to curated urban soundscapes, using the same equipment and technical specifications as all other intervention conditions. Each participant is randomly assigned one of 22 recordings, calibrated to 60-70 dB (Leq,20min). The recordings feature anthropophony (e.g., unintelligible background speech) and technophony (e.g., transportation-related sounds), free of natural sounds and selected for ecological validity based on the same predefined criteria as the natural soundscapes. To prevent semantic processing, participants are pre-screened and post-session reconfirmed to ensure they do not understand the languages used. During exposure, participants lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening and is conducted under continuous researcher supervision.
  Other Names: Experimental intervention U
Other: Broadband sound exposure — Participants receive a standardized 20-minute auditory exposure to broadband sounds (i.e., white or pink noise), using the same equipment and technical specifications as all other intervention conditions. Each participant is randomly assigned to one of the two noise types, with equal distribution across conditions. The stimuli are generated using professional audio software and calibrated to 50 dB (Leq,20min). During exposure, participants lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening and is conducted under continuous researcher supervision.
  Other Names: Active comparator
Other: Blank tape attention placebo control — Participants receive a standardized 20-minute exposure to blank audio (silence), using the same equipment and technical specifications as all other intervention conditions. At study onset, participants are informed they will hear a range of environmental sounds, including some that may be inaudible (i.e., present but beyond the range of human hearing). During the placebo condition, a blank recording is played, producing silence, while participants remain unaware of whether they are receiving an active or placebo stimulus. This attention-control condition ensures procedural consistency while delivering no auditory stimulation. During exposure, participants lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening and is conducted under continuous researcher supervision.
  Other Names: Placebo comparator

SUMMARY:
This study examines whether different types of sounds can help reduce pain in people with fibromyalgia, a chronic condition that causes widespread pain and increased sensitivity to sensory experiences. Fibromyalgia affects approximately 2-3% of the global population and has limited treatment options. Recent research suggests that environmental sounds might have the capacity to influence pain perception, but their effects in chronic pain conditions remain largely unexplored. Such research could lead to new, non-invasive, sound-based approaches for managing fibromyalgia pain and inform the design of healthier acoustic environments for people with chronic pain conditions.

The study will compare four different sound environments: natural soundscapes (like birdsong and rainfall), urban soundscapes (like traffic and background conversation), broadband sounds (white or pink noise), and silence (as a neutral/control condition with intended placebo effect). Researchers want to know if these different sound environments can change how people with fibromyalgia experience pain and if some environmental sounds might be more helpful than others.

Each participant will experience all four sound conditions in a random order, with one session per week over four weeks. With this study design, each participant acts as their own control, which reduces differences between individuals and increases the reliability of the results. During each 20-minute session, participants will listen to the assigned sounds through a high-fidelity sound reproduction setup using headphones while lying comfortably on a padded therapy table in a controlled laboratory setting. Before and after each sound exposure, researchers measure pain intensity and sensitivity using standardized assessments to determine whether and how different sound environments, if any, might offer pain relief.

DETAILED DESCRIPTION:
This protocol investigates the potential modulatory effects of distinct auditory environments on pain processing mechanisms in individuals with fibromyalgia syndrome. The study is grounded in emerging neuroscientific evidence suggesting that auditory stimuli can influence pain perception through direct neural pathways between the auditory cortex and pain-processing regions.

Soundscapes-defined as acoustic environments perceived, experienced, and interpreted within specific contexts-are categorized as natural or anthropogenic based on their origin for research purposes. Natural soundscapes comprise elements such as biophonies (non-human animal sounds) and geophonies (non-living natural elements), while urban soundscapes feature anthropophonies (human-generated sounds) and technophonies (mechanical sources). Recent neuroimaging research has demonstrated that these different soundscape categories elicit distinct neural signatures and may differentially shape intrinsic brain dynamics.

Fibromyalgia syndrome presents a particularly relevant clinical model for investigating auditory-pain interactions due to its characteristic heightened sensitivity to non-noxious sensory input. Preclinical evidence has identified direct neural pathways between the auditory cortex and pain-processing regions, with rodent studies showing that 20-minute broadband sound exposure significantly increases mechanical pain thresholds through mechanisms involving reduced thalamic activity. Human studies have similarly documented analgesic effects of auditory stimulation across both acute experimental pain and chronic pain conditions.

The general objective of this study is to:

GO1. Investigate the differential effects of controlled auditory environmental exposures-natural soundscapes, urban soundscapes, broadband sound, and silence-on the functioning of altered pain mechanisms in individuals with fibromyalgia syndrome, evaluated through clinical outcomes (pain intensity and perceived improvement) and experimental indices of pain processing (quantitative sensory testing measures).

The specific objectives are to:

SO1. Compare the effects of natural and urban soundscapes against broadband sound (active comparator) and silence (attention-placebo control) on the functioning of pain mechanisms.

SO2. Determine the relative efficacy of natural versus urban soundscapes in modulating the functioning of pain mechanisms in individuals with fibromyalgia syndrome.

SO3. Characterize the magnitude and direction of potential within-condition changes in the functioning of pain mechanisms following exposure to natural and urban soundscapes.

The primary hypothesis is:

PH1. Distinct auditory environmental exposures-natural soundscapes, urban soundscapes, broadband sound, and silence-will differentially modulate self-reported pain intensity in individuals with fibromyalgia syndrome, with the following specific hypothesized relationships:

PH1.1. Natural soundscape exposure will demonstrate superior analgesic efficacy compared to attention-placebo control.

PH1.2. Natural soundscape exposure will demonstrate superior analgesic efficacy compared to broadband sound exposure.

PH1.3. The analgesic effects of urban soundscape exposure will not significantly differ from attention-placebo control.

PH1.4. The analgesic effects of urban soundscape exposure will not significantly differ from broadband sound exposure.

PH1.5. Natural soundscape exposure will demonstrate superior analgesic efficacy compared to urban soundscape exposure.

The secondary hypotheses are:

SH1. Exposure to natural soundscapes will lead to significant pre-post improvements in both clinical outcomes and experimental indices of pain processing.

SH2. Exposure to urban soundscapes will demonstrate non-significant pre-post effects in both clinical outcomes and experimental indices of pain processing.

The study design optimizes statistical efficiency by allowing within-subject comparisons while controlling for period effects. The auditory exposure sessions are conducted in a controlled laboratory environment, maintaining a consistent room temperature and relative humidity.

To recruit participants, voluntary response, convenience, and snowball sampling methods will be employed. An a priori power analysis was conducted using G*Power v3.1.9.7. The sample size estimation is based on a Cohen's f effect size of 0.516, derived from the previous findings on the effect of nature sounds on pain in patients with chronic pain. A minimum of 58 participants is required to provide a power of 90% to adequately detect the determined pre-post difference at a two-tailed alpha level of .05. Allowing for an anticipated attrition rate of approximately one-third-including potential dropout, loss to follow-up, clinical reasons, and operational issues-a total of 88 participants will be recruited.

The assessment protocol follows International Association for the Study of Pain consensus guidelines and incorporates core outcome domains recommended for chronic pain trials. It covers both clinical outcomes (pain intensity and perceived improvement) and experimental indices of pain processing (quantitative sensory testing measures). These measures collectively provide a comprehensive evaluation of both subjective pain experience and biomarkers of pain processing, performed by a trained evaluator.

The primary analytical strategy will use linear mixed-effects models to examine change-from-baseline scores across conditions. Fixed effects will include treatment, period, sequence, and their interaction to detect potential carryover effects, while participants will be modeled with random intercepts. In the absence of carryover, a simplified model excluding the interaction term will be applied. Between-condition effects will be assessed via estimated marginal means with Bonferroni-adjusted pairwise comparisons. Sensitivity analyses will introduce the covariates to examine their influence on treatment effects. Within-condition (pre-post) changes will be evaluated using paired t-tests or Wilcoxon signed-rank tests, depending on data distribution.

To meet statistical assumptions, distributions of quantitative sensory testing outcomes-including mechanical pain sensitivity, temporal summation of pain, and pressure pain detection thresholds and intensity ratings-will be log-transformed, consistent with established methods. A small constant will be added to variables with potential zero values prior to transformation. For presentation purposes, transformed values will be back-converted to original units in descriptive outputs. All hypothesis testing will be two-sided with a Type I error rate of 5%, and analyses will follow the intention-to-treat principle. Multiple imputation will be considered if missingness is not at random.

This study is considered as minimal risk. No serious adverse events are expected. All participants may withdraw at any time without justification or impact on healthcare access. Discontinuation may occur at participants' request or in response to adverse events or protocol violations. Adverse events will be monitored throughout. Given the low-risk profile, oversight will be managed by the principal investigator; no independent safety board is planned. Safety monitoring will involve systematic documentation of all treatment-emergent and spontaneously reported adverse events throughout the study period.

To our knowledge, this study would represent one of the first investigations conceptualizing everyday soundscapes as environmental determinants potentially capable of modulating pain processing in chronic pain populations. The findings may contribute to several domains:

1. Theoretical advancement in understanding auditory-pain interactions and their environmental influences.
2. Development of novel, non-pharmacological auditory-based interventions for pain management in fibromyalgia syndrome.
3. Informing environmental health policies and acoustic design strategies for healthcare settings.
4. Contributing to the emerging field of environmental neuroscience by informing whether and how environmental sounds influence chronic pain processing.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of fibromyalgia syndrome, documented in the medical record provided by the participant prior to enrollment.
* Moderate or greater pain intensity during the preceding week, defined as a score higher than 3 on an 11-point Numeric Rating Scale.
* Normal hearing confirmed by a hearing test, defined as a mean threshold of ≤ 20 dB HL at 0.125, 0.25, 0.5, 1, 2, 4, 6, and 8 kHz.
* Ability to communicate in Spanish.
* Provision of signed written informed consent to participate in the research.

Exclusion Criteria:

* A diagnosis of misophonia or auditory processing disorders, as documented in the participant's medical record.
* Concurrent neuropathic or acute pain.
* Severe cognitive impairment, defined as a Mini-Mental State Examination score ≤ 17.
* Severe psychiatric disorders in the symptomatic phase.
* History of substance abuse in the past 12 months or current substance use disorder as reported by the participant.
* Changes in ongoing therapy during or within one month prior to study enrollment per participant self-reports.
* Central nervous system disorders.
* Any other serious or unstable medical condition that could interfere with study participation.
* Known allergies or hypersensitivity to study materials.
* Pregnancy, lactation, or being within three months postpartum at the time of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from immediately before to immediately after each 20-minute intervention session during each of the four crossover periods
  The primary outcome measure assesses acute changes in subjective pain intensity following each auditory intervention. Participants mark their current pain level on a 100-mm Visual Analog Scale anchored from "no pain" to "the worst pain imaginable". The scale is scored as the distance in millimeters from the left end, with lower scores corresponding to lower perceived pain.

SECONDARY OUTCOMES:
Patient global impression of change | Assessed immediately after each 20-minute intervention session during each of the four crossover periods
  Participants rate overall change on a seven-point Likert scale ranging from one ("very much improved") to seven ("very much worse"). Lower scores indicate greater perceived improvement.
Mechanical pain sensitivity | Change from immediately before to immediately after each 20-minute intervention session during each of the four crossover periods
  Mechanical pain sensitivity is assessed using a response-dependent procedure with a 180-gram Semmes-Weinstein monofilament, involving three perpendicular stimulations to the cheek on each side, with 10-second interstimulus intervals. After each application, participants rate the perceived pain intensity on a 100-mm Visual Analog Scale. This sequence is repeated three times, and the geometric mean of the three ratings is calculated for each side. The arithmetic mean of the bilateral geometric means is registered as the mechanical pain sensitivity. Lower values indicate lower mechanical pain sensitivity.
Temporal summation of pain | Change from immediately before to immediately after each 20-minute intervention session during each of the four crossover periods
  Temporal summation is assessed using a response-dependent procedure with a 180-gram Semmes-Weinstein monofilament applied to the left thenar eminence. First, a single stimulus is administered, followed by participant rating of perceived pain intensity on a 100-mm Visual Analog Scale. After a 30-second interval, a series of 10 stimuli is delivered at 1 Hz to the same location, followed by an overall pain rating. The temporal summation index is calculated as the difference between the pain ratings for the stimulus series and the single stimulus. Lower values indicate reduced central pain facilitation.
Pressure pain detection thresholds and intensity ratings | Change from immediately before to immediately after each 20-minute intervention session during each of the four crossover periods
  Pressure pain detection thresholds are assessed using a digital pressure algometer equipped with a one-cm² circular flat probe, following the method of limits. Assessment sites include the midpoint of the upper trapezius and the medial fat pad of the knee, measured bilaterally. Pressure is applied at a constant rate of 50 kPa/sec until participants report the first perception of pain, with a maximum cutoff of 1000 kPa for safety. Three trials are performed per site, with the first trial discarded. The arithmetic mean of the second and third trials across all four sites is recorded as the pressure pain threshold. Following each application, participants rate the evoked pain intensity using a 100-mm Visual Analog Scale. The mean of the second and third intensity ratings across all sites is registered as the pressure-evoked pain intensity. Higher threshold values indicate lower pain sensitivity, while lower intensity scores reflect reduced perceived pain.

OTHER OUTCOMES:
Somatosensory amplification | Assessed at baseline
  The Somatosensory Amplification Scale evaluates the extent to which individuals perceive normal bodily sensations as exaggerated or disturbing, across two dimensions: internal and external amplification. It includes 10 items rated on a five-point Likert scale, ranging from one ("not at all") to five ("extremely"), yielding a total score of 10-50. Higher scores reflect greater somatosensory amplification.
Pain catastrophizing | Assessed at baseline
  The Pain Catastrophizing Scale evaluates participants' tendency to catastrophize pain. It consists of 13 items across three dimensions-rumination, magnification, and helplessness-rated on a five-point Likert scale, ranging from zero ("not at all") to four ("all the time"). Total scores range from 0 to 65, with higher values indicating greater catastrophizing.
Connectedness to nature | Assessed immediately after the final 20-minute intervention session, following completion of all other outcome assessments during the fourth crossover period (Week 4)
  The Connectedness to Nature Scale assesses participants' attitudes toward nature. The self-report scale comprises 13 items rated on a five-point Likert scale, ranging from one ("strongly disagree") to five ("strongly agree"). The total score ranges from 13 to 65, with higher scores reflecting a greater sense of connectedness to nature.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Pérez Mármol, PhD, Principal Investigator — Department of Physiotherapy, Faculty of Health Sciences, University of Granada
Locations (1):
- Faculty of Health Sciences, University of Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be shared after de-identification, in accordance with executed data sharing agreements that require adherence to confidentiality, data protection, and non-reidentification standards equivalent to those of the originating study. The data to be shared will include baseline participant characteristics, outcome measures, covariates, and safety data. Only data necessary to replicate study findings or to conduct methodologically sound secondary analyses will be made available. The shared dataset will be accompanied by a comprehensive data dictionary that defines all variables, coding schemes, and measurement protocols to ensure full interpretation and appropriate use of the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests may be submitted beginning 12 months after the article's publication. The data will remain available for up to 24 months thereafter. Requests for extended access will be considered on a case-by-case basis and may be granted if appropriately justified.
Access Criteria: Data will be shared with qualified researchers who submit a methodologically sound proposal for analyses that align with the aims outlined in the approved application. Proposals should demonstrate scientific merit, methodological rigor, and the potential to advance understanding of chronic pain or auditory interventions. Requestors must sign a data sharing agreement that includes commitments to use the data only for approved purposes, implement appropriate data security measures, acknowledge the original study in any resulting publications, and share results with the original research team. For additional details or to initiate a request, please contact josemapm@ugr.es